CLINICAL TRIAL: NCT05189392
Title: Effect of PICO Compared to Opsite Post-Op Visible on Surgical Wound in Patients at High Risk of Local Complications, Undergoing Hip Arthroplasty
Brief Title: Efficacy of PICO Compared to Opsite Post-Op Visible on Surgical Wound in Patients at High Risk of Local Complications, Undergoing Hip Arthroplasty
Acronym: PICO-PTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICO-PTA
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Evaluate Postsurgical Hematoma

STUDY DESIGN:
Intervention Model Description: 21 patients with visible opsite patch and 21 patients with PICO
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 21 patients with opsite visible (No Intervention): application of visible opsite plaster on the surgical wound after hip arthroplasty
- 21 patients with PICO (Experimental): application of PICO on the surgical wound after hip arthroplasty
  Interventions: Device: PICO

INTERVENTIONS:
Device: PICO — after hip arthroplasty application of visible opsite plaster on the surgical wound
  Other Names: Opsite Visible
  Arms: 21 patients with PICO

SUMMARY:
Evaluate the effect of the PICO medical device, compared to the Opsite Post-Op Visible medical device, in reducing the formation of postsurgical hematoma in the surgical wound of patients at high risk of local complications, undergoing hip arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* aged between 55 and 85 years inclusive,
* Patients with BMI ≥ 30 + ASA 3 + Diabetes mellitus
* Patients suffering from coxarthrosis candidates for hip arthroplasty surgery or revision of hip arthroplasty

Exclusion Criteria:

* Age> 85 years, <55 years
* Patients who are unable to understand and want.
* Patients with severe neurological disorders or with severe disabilities.
* Oncological patients and patients with malignant tumor at the edge of the wound
* Patients who have undergone radiotherapy treatment
* Patients with bleeding disorders
* Patients on anticoagulant treatment with warfarin or NAO
* Previously confirmed osteomyelitis
* Patients with liver cirrhosis
* Patients with non-enteric fistulas
* Patients with necrotic tissue with the presence of eschar at the intervention site
* Patients with autoimmune thrombocytopenia.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
By ultrasound examination at 7 +/- 1 days after hip replacement surgery, underestimating the effect of PICO compared to Opsite Post-Op Visible in the 70% reduction of post-surgical hematoma formation | 8 day
  By ultrasound examination at 7 +/- 1 days after hip replacement surgery, underestimating the effect of PICO compared to Opsite Post-Op Visible in the 70% reduction of post-surgical hematoma formation

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, MI, Italy